CLINICAL TRIAL: NCT01175200
Title: Double the Dose of Clopidogrel or Switch to Prasugrel to Antagonize Proton Pump Inhibitor Interaction. A Prospective, Mono-center, Placebo- and Active Treatment-controlled, Randomized, Cross Over Study.
Brief Title: Double the Dose of Clopidogrel or Switch to Prasugrel to Antagonize Proton Pump Inhibitor Interaction.
Acronym: DOSAPI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ascopharm Groupe Novasco (Other)
Collaborators: Groupe Hospitalier Pitie-Salpetriere (Other); Medco Health Solutions, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DOSAPI
Record Dates: First submitted 2010-08-03; First posted 2010-08-04 (Estimated); Last update posted 2012-07-04 (Estimated); Status verified 2012-07

CONDITIONS: Anti Platelet Effects
MeSH Terms: interventions — Clopidogrel; Prasugrel Hydrochloride; Lansoprazole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Prasugrel (Active Comparator)
  Interventions: Drug: Prasugrel
- Clopidogrel (Active Comparator)
  Interventions: Drug: Clopidogrel
- Lansoprazole (Active Comparator): proton pump inhibitor
  Interventions: Drug: Lansoprazole
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Clopidogrel — antiplatelet agent
  Arms: Clopidogrel
Drug: Prasugrel — antiplatelet agent
  Arms: Prasugrel
Drug: Lansoprazole — proton pum inhibitor
  Other Names: Lanzor; Ogast
  Arms: Lansoprazole
Drug: Placebo — placebo comparator similar to lansoprazole
  Arms: Placebo

SUMMARY:
This study will establish the optimal therapeutic strategy for patients with a coronary artery disease (CAD) and chronically treated with clopidogrel 75 mg/day requiring co-administration of an anti-platelet treatment with P2Y12 antagonist and a PPI for treatment/prevention of GI ulceration.

ELIGIBILITY:
Inclusion Criteria :

* patient with stable Coronary Artery Disease (< 3 months) treated with clopidogrel (75mg/d)
* Between 18 and 75 years of age
* Body Mass Index between 18 and 30 kg/m2 and body weight not less than 60 kg
* No major bleeding according to ISTH definition
* Subjects who signed an informed consent document
* Subjects who signed a separate pharmacogenomic informed consent document
* Subjects registered to the French national welfare system

Exclusion Criteria:

* Personal or family history of coagulation or bleeding disorders
* Use of known inhibitors or inducers of CYP2C19 and CYP3A including grape fruit juice intake
* Known hypersensitivity to lansoprazole, its excipients, or substituted benzimidazoles,
* Known hypersensitivity to clopidogrel / prasugrel
* Anti-platelet treatment other than clopidogrel + aspirin within 7 days before inclusion
* Any formal indication to maintain PPI treatment
* PPI within 15 days before inclusion in the study
* Active pathology with 10 days before inclusion
* Prior history of stent thrombosis
* Prior history of Stroke
* Employee of the investigator or study center, with direct involvement in the proposed study or other studies under the direction of that investigator or study center, as well as family members of the employees or the investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2010-09; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Change in antiplatelet effect of clopidogrel | 14 days
  change in antiplatetelet effect of clopidogrel as compared to prasugrel when associated to lansoprazole (or placebo) in patients with stable angina

SECONDARY OUTCOMES:
high on-treatment platelet reactivity Clopidogrel pharmacokinetics responses | 14 days
  compare persistant antiplatelet hyper reactivity in patients with stable angina and treated with clopidogrel or prasugrel associated with lansoprazole (or placebo)

CONTACTS AND LOCATIONS:
Locations (1):
- Pitié Salpétrière Hospital, Paris, France